CLINICAL TRIAL: NCT06932068
Title: Safety and Efficacy of Iparomlimab and Tuvonralimab (QL1706) Combined With Chemotherapy for the Treatment of HER2-Negative, Low PD-L1 Expressing, Unresectable or Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma: A Phase II Single-Arm Trial
Brief Title: Phase II Trial of Iparomlimab/Tuvonralimab (QL1706) + XELOX in HER2-Negative, Low PD-L1 G/GEJ Adenocarcinoma
Acronym: SEARCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Lian Liu, MD, PHD, Director of Department of Oncology, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEARCH
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: HER2 Negative; Low PD-L1 Expressing; Unresectable or Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 + XELOX chemotherapy (Experimental): Iparomlimab and Tuvonralimab+XELOX
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706); Drug: Oxallplation; Drug: Capectitabine Tablets

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab (QL1706) — 5 mg/kg, ivdrip, Day 1, Q3W, until progressive disease or intolerable toxicity.
Drug: Oxallplation — 130 mg/m2, ivdrip, Day 1, Q3W, for the first 6 cycles.
Drug: Capectitabine Tablets — 1000 mg/m2, po, bid, Days 1-14, Q3W, until progressive disease or intolerable toxicity.

SUMMARY:
This is single - arm study to explore the safety and efficacy of iparomlimab and tuvonralimab (QL1706) combined with chemotherapy for treating her2-negative, low PD-L1 expressing, unresectable or metastatic gastric/gastroesophageal junction adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, gender is not limited;
2. Pathologically confirmed locally advanced gastric or gastroesophageal junction adenocarcinoma that is inoperable or has distant metastasis;
3. HER2-negative by immunohistochemistry (IHC);
4. low PD-L1 expression status (CPS < 5);
5. Has at least 1 measurable lesion as determined by RECIST 1.1;
6. No systematic treatment in the past, or the patient has received neoadjuvant/adjuvant chemotherapy, but the disease progresses or relapses more than 6 months after the end of treatment;
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
8. Adequate organ function;
9. The life expectancy is at least 3 months;
10. Willing to join the study and signed an informed consent form (ICF) with good compliance and cooperation in follow-up.

Exclusion Criteria:

1. Allergic to any trial drug and its excipients, or serious allergy history, or contraindication of the trial drug;
2. Cardiovascular and cerebrovascular events that are not well controlled;
3. Has received systematic treatment with Chinese patent medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use for ascites control) before the first administration within 2 weeks;
4. Have a history of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, acute lung disease, or systemic disease with poor control (including but not limited to diabetes, hypertension, etc.);
5. Have a history of active immune deficiency or autoimmune diseases, including HIV positive test, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation or autoimmune diseases;
6. Severe chronic or active infection requires systemic antibacterial, antifungal or antiviral treatment, including tuberculosis infection.Have a history of active tuberculosis infection ≥ 1 year before recruitment should also be excluded, unless proved has been completed appropriate treatment;
7. Brain metastasis or leptomeningeal metastasis;
8. Clinically significant pleural effusion, pericardial effusion or ascites should be drained for many times within 2 weeks before the first administration of the trial drug;
9. Has a second clinically detectable primary malignant tumor at the time of recruitment, or there were other malignant tumors in the past 5 years (except for fully treated skin basal cell carcinoma or cervical carcinoma in situ);
10. Any major surgery was performed ≤ 28 days before the first trial drug administration;
11. History of allogeneic stem cell transplantation or organ transplantation;
12. Duodenal ulcer, ulcerative colitis, intestinal obstruction and other gastrointestinal diseases at present; or other conditions that may cause gastrointestinal bleeding or perforation judged by the researchers; or history of intestinal perforation or fistula, but has not recovered after surgical treatment;
13. Live vaccine was inoculated within 4 weeks (inclusive) before the first administration of the trial drug, not including seasonal influenza vaccines but intranasal vaccine.
14. Has other factors that may lead to the forced termination of this trial according to the judgment of the investigator, such as other serious diseases (including psychological and mental diseases) requiring combined treatment, serious laboratory examination abnormalities, and family or social factors, which may affect the safety of the subject, or the collection of data and samples;
15. Participating in other therapeutic clinical studies or using research instruments within 4 weeks before the first administration;
16. Others conditions do not meet the inclusion according to the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 12 months after the last subject participating in
  The time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first (per RECIST 1.1).

SECONDARY OUTCOMES:
overall survival (OS) | 12 months after the last subject participating in
  The time from the starting date of study drug to the date of death due to any cause.
objective response rate (ORR) | 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) according RESIST1.1 in total subjects.
duration of response (DOR) | 12 months after the last subject participating in
  The time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
disease control rate (DCR) | 12 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease(SD) in total subjects
Safety (adverse event) | Up to approximately 2 years
  The rates of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Liu, MD, PHD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided